CLINICAL TRIAL: NCT02944682
Title: Household Air Pollution and Health: A Multi-country LPG Intervention Trial
Acronym: HAPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Bill and Melinda Gates Foundation (Other); Berkeley Air Monitoring Group (Other); Colorado State University (Other); Global LPG Partnership (Unknown); Harvard University (Other); Johns Hopkins University (Other); London School of Hygiene and Tropical Medicine (Other); Asociacion Benefica Prisma (Other); Sri Ramachandra University (Other); Universidad del Valle, Guatemala (Other); Universidad Peruana Cayetano Heredia (Other); University of Georgia (Other); Washington University School of Medicine (Other); University of Rwanda (Other); Eagle Research Center (Unknown); University of Oxford (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Thomas Clasen, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00089799; 1UM1HL134590-01 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-26 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Infant, Low Birth Weight
Keywords: Obstetrics; Pregnancy Outcomes; Pediatrics; Atherosclerosis; Cancer; Cardiovascular Disease; Public Health; Environmental Air Pollutants
MeSH Terms: conditions — Atherosclerosis; Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquefied petroleum gas cookstove (Experimental): Participants randomized to the experimental arm will receive a liquefied petroleum gas (LPG) cookstove and 18-month supply of LPG.
  Interventions: Other: Liquefied petroleum gas (LPG) cookstove
- Control (No Intervention): Participants in the control group will not receive a liquefied petroleum gas (LPG) stove and will continue using traditional cooking methods (open fire or traditional stoves), or the cooking method of their choice. Control households will receive compensation based on a uniform set of trial-wide principles, customized to each site based on formative research.

INTERVENTIONS:
Other: Liquefied petroleum gas (LPG) cookstove — The intervention consists of a high-quality locally-available liquefied petroleum gas (LPG) stove having at least two burners, a continuous supply of LPG fuel for 18 months, and the promotion of stove use on an exclusive basis for cooking. The intervention will be provided free of charge to all intervention households upon enrollment. On a weekly basis, study staff will examine stove condition, perform any repairs necessary, and measure and record weight of LPG tanks in order to anticipate need for refills.
  Arms: Liquefied petroleum gas cookstove

SUMMARY:
This study is a randomized controlled trial of liquefied petroleum gas (LPG) stove and fuel distribution in 3,200 households in four countries (India, Guatemala, Peru, and Rwanda). Following a common protocol, each intervention site will recruit 800 pregnant women (aged 18-34 years, 9 - <20 weeks gestation), and will randomly assign half their households to receive LPG stoves and an 18-month supply of LPG. Control households are anticipated to continue to cook primarily with solid biomass fuels, and will receive compensation based on a uniform set of trial-wide principles, customized to each site based on formative research. The mother will be followed along with her child until the child is 1 year old. The researchers estimate that 15% of households will have a second, non-pregnant older adult woman (aged 40 to <80 years) who will also be enrolled at baseline and followed during the 18-month follow-up period. To optimize intervention use, the researchers will implement behavior change strategies informed by previous experiences and formative research in Year 1. This study will assess cookstove use, conduct repeated personal exposure assessments of household air pollution, and collect dried blood spots and urinary samples for biomarker analysis and biospecimen storage. The primary outcomes are low birth weight, severe pneumonia incidence, and stunting of the child, and systolic blood pressure in the older adult woman. Participants in India, Guatemala and Rwanda will be followed until the child is 5 years old to assess the longer-term effects of the intervention.

DETAILED DESCRIPTION:
Globally, nearly 3 billion people rely on solid fuels for cooking and heating, the vast majority in low- and middle-income countries (LMICs). The resulting household air pollution (HAP) is the third leading risk factor in the 2010 global burden of disease, accounting for an estimated 4.3 million deaths annually, largely among women and young children. Previous interventions have provided cleaner biomass-based cookstoves, but have failed to reduce exposure to levels that produce meaningful health improvements. There have been no large-scale field trials with liquefied petroleum gas (LPG) cookstoves, likely the cleanest scalable intervention.

The aim of this study is to conduct a randomized controlled trial of LPG stove and fuel distribution in 3,200 households in four LMICs (India, Guatemala, Peru, and Rwanda) to deliver rigorous evidence regarding potential health benefits across the lifespan. Each intervention site will recruit 800 pregnant women (aged 18-34 years, 9 - <20 weeks gestation), and will randomly assign half their households to receive LPG stoves and an 18-month supply of LPG. Control households are anticipated to continue to cook primarily with solid biomass fuels, and will receive compensation based on a uniform set of trial-wide principles, customized to each site based on formative research. The mother will be followed along with her child until the child is 1 year old. In households with a second, non-pregnant older adult woman (aged 40 to <80 years) the researchers will also enroll and follow her during the 18-month follow-up period in order to assess cardiopulmonary, metabolic, and cancer outcomes. To optimize intervention use, the researchers will implement behavior change strategies. This study will assess cookstove use, conduct repeated personal exposure assessments to HAP (PM2.5, black carbon, carbon monoxide), and collect dried blood spots and urinary samples for biomarker analysis and biospecimen storage on all participants at multiple time points. The primary outcomes are low birth weight, severe pneumonia incidence, and stunting of the child, and systolic blood pressure in the older adult woman.

This study will address the following specific aims: (1) using an intent-to-treat analysis, determine the effect of a randomized LPG stove and fuel intervention on health in four diverse LMIC populations using a common protocol; (2) determine the exposure-response relationships for HAP and health outcomes; and (3) determine relationships between LPG intervention and both targeted and exploratory biomarkers of exposure/health effects.

This study will provide evidence, including costs and implementation strategies, to inform national and global policies on scaling up LPG stoves among vulnerable populations. Ultimately, this will facilitate deeper policy-level discussions as well as identify requirements for initiating and sustaining HAP interventions globally.

The intervention delivery occurred until the child was one year of age. The researchers will continue to follow participants in India, Guatemala and Rwanda until the child is 5 years old to assess the longer-term effects of the intervention. Previous evidence suggests that the benefits of reduced exposure during the first, critical year of development will continue even if the intervention ends. The researchers will continue using methods employed during the HAPIN trial period. The HAPIN trial provides a unique context in which to address these questions, particularly given the successful intervention and exposure reduction. Participants are well-characterized and health and exposures to air pollution are being documented. Critically, because of its experimental design of the trial, continued follow-up of the cohort will provide rigorous causal inferences about the effects of this 500-day intervention over the most important period of early childhood development.

ELIGIBILITY:
Inclusion Criteria for Pregnant Women:

* Confirmed pregnancy (hCG positive blood or urine test)
* Aged 18 to <35 years (via self-report)
* Uses biomass stove predominantly
* Lives in study area
* 9 - <20 weeks gestation confirmed by ultrasound
* Singleton pregnancy (one fetus)
* Viable fetus with normal fetal heart rate (120-180 beats per minute) at time of ultrasound
* Continued pregnancy at the time of randomization confirmed by self-report
* Agrees to participate with informed consent

Exclusion Criteria for Pregnant Women:

* Currently smokes cigarettes or other tobacco products
* Plans to move permanently outside study area in the next 12 months
* Uses LPG stove predominantly, or is likely to use LPG predominantly in the near future

Inclusion Criteria for Older Adult Woman in the Same Household:

* Aged 40 to <80 years (via self-report)

Exclusion Criteria for Older Adult Woman in the Same Household:

* Currently smokes cigarettes or other tobacco products
* Pregnant (by self-report)
* Plans to move out of her current household in the next 12 months

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3640 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Birth weight | Within 24 hours of birth (up to 5 months post-randomization of mother)
  Birth weight will be assessed by a trained nurse or health worker within 24 hours of birth. Infants will be weighed naked or in a pre-weighed blanket. Weight will be measured to the nearest 10 g using a digital electronic scale, if performed by the study field staff; otherwise, hospital medical records will be used.
Incidence of HAPIN Defined Severe Pneumonia | Up to 12 months after birth
  The number of times a child has severe pneumonia over their period of follow-up during the first year of life will be assessed. HAPIN pneumonia criteria are adapted from the WHO classification of childhood pneumonia (2014) and there are 3 algorithms for HAPIN case criteria: 1) the presence of cough and/or difficult breathing and at least 1 general danger sign plus evidence of pneumonia on lung imaging (i.e., lung ultrasound or chest x-ray), or 2) the presence of cough and/or difficult breathing and hypoxemia (measured either via pulse oximetry (SpO2), or observing a child requiring advanced respiratory support (i.e., intubation and mechanical ventilation, non-invasive ventilation with continuous or bi-level positive airway pressure support, or high-flow nasal cannula oxygen), or 3) children who die prior to evaluation but their death is attributed to pneumonia by verbal autopsy. Cases of pneumonia are recorded children present to HAPIN health facilities with respiratory symptoms.
Length-for-age z-score 2 standard deviations below the standard | 12 months after birth
  The primary outcome measured is stunting at one year of age, defined as a length-for-age z-score (LAZ) that is 2 standard deviations below the median of the growth standard. Infant length will be assessed at birth and quarterly thereafter, until the child is 12 months old. Z-scores will be calculated using the 2006 World Health Organization (WHO) Multi-Growth Reference Standard (MGRS).
Change in Systolic Blood Pressure | Baseline, 3, 5, 9, 12, and 18 months post-randomization (24, 36, 48, and 60 months of age)
  Systolic blood pressure will be assessed in the older adult women in the intervention and control arms using automatic sphygmomanometers (Omron HEM-907XL; Osaka, Japan). The study team will use the procedures adapted from previously validated methods and cardiovascular outcome studies, following recommendations for the American Heart Association and the European Society of Hypertension.
Change in Child Linear Growth | Birth (3-5 months post-randomization), and 3, 6, 9, 12, 24, 36, 48 and 60 months of age
  Linear growth of children will be assessed in centimeters of height from the time of birth until 60 months of age.
Change in Caregiver Reported Early Childhood Development Instrument (CREDI) Score | 3 months of age to 24 months of age
  Child development will be assessed with the Caregiver Reported Early Childhood Development Instrument (CREDI). The CREDI is a population-level measure of early childhood development (ECD) for children from 0-2 years of age. The CREDI assesses 5 domains of child development: 1) motor development (fine and gross motor), 2) language development (expressive and receptive language), 3) cognitive development (executive function, problem solving and reasoning, and pre-academic knowledge), 4) socio-emotional development (emotional and behavioral self-regulation, emotional knowledge, and social competence), and 5) mental health (internalizing and externalizing behaviors). The CREDI long form has 117 items and the number of questions answered depends on the age of the child. Responses of "yes" are coded as 1 and "no" is coded as 0; certain items are reverse coded. Total raw scores increase by age (with developmental progression), and higher scores indicate increased development.
Change in Malawi Developmental Assessment Tool (MDAT) Score | 36, 48 and 60 months of age
  The MDAT measures gross motor (39 items), fine motor (42 items), language/cognition (40 items) and social skills (36 items). Originally developed and validated in rural Malawi, it has now been used in over 25 countries with more than 8,000 children as both a clinical and research tool. The MDAT is a continuous test with start and stop rules. Most items are administered directly to the child and items that are not easily observed (e.g., child speaks in full sentences; child understands sharing with others; child can dress self) are administered by parent report. Children receive either a pass or fail for each item, and summed pass scores can produce a composite score as well as domain-specific scores. Total scores range from 0 to 157 where higher scores indicate greater neurodevelopment.

SECONDARY OUTCOMES:
Change in Maternal Blood Pressure | Baseline (9-20 weeks gestation), 24-28 and 32-36 weeks gestation, and at 24, 36, 48 and 60 months of age of the child
  Blood pressure will be assessed in the pregnant women in the intervention and control arms using automatic sphygmomanometers (OMRON HEM-907XL; Osaka, Japan). After delivery, blood pressure will be measured in the new mothers when the child is 24, 36, 48 and 60 months old. The study team will use the procedures adapted from previously validated methods and cardiovascular outcome studies, following recommendations for the American Heart Association and the European Society of Hypertension.
Change in Diastolic blood pressure | Baseline, 3, 6, 12 and 18 months post-randomization, and at 24, 36, 48, and 60 months of age of the child
  Diastolic blood pressure will be assessed in the older adult women and new mothers in the intervention and control arms using automatic sphygmomanometers (Omron HEM-907XL; Osaka, Japan). The study team will use the procedures adapted from previously validated methods and cardiovascular outcome studies, following recommendations for the American Heart Association and the European Society of Hypertension.
Mean arterial pressure | Baseline, 3, 6, 12 and 18 months post-randomization, and at 24, 36, 48, and 60 months of age of the child
  Mean arterial pressure will be assessed in the older adult women and new mothers in the intervention and control arms using automatic sphygmomanometers (Omron HEM-907XL; Osaka, Japan). Mean arterial pressure is calculated as DBP+(SBP-DBP)/3, where SBP=systolic blood pressure and DBP=diastolic blood pressure.
Pulse pressure | Baseline, 3, 6, 12 and 18 months post-randomization, and at 24, 36, 48, and 60 months of age of the child
  Pulse pressure will be assessed in the older adult women and new mothers in the intervention and control arms using automatic sphygmomanometers (Omron HEM-907XL; Osaka, Japan). pressure. Pulse pressure is the difference between systolic blood pressure and diastolic blood pressure.
Fetal Growth | Baseline, Gestation Week 24-28 and Gestation Week 32-36
  Pregnant women will have ultrasounds at Baseline and during gestation weeks 24-28 and gestation weeks 32-36 to measure fetal growth outcomes. Specifically, we will evaluate head circumference (HC), abdominal circumference (AC), femur length (FL) and estimated fetal weight (EFW) during gestation. We will compare (i) z-scores of individual fetal growth measurements (HC, AC, FL, EFW) at the 2 growth ultrasound visits between intervention and control participants (separately at 24-28 wks gestation and 32-36 wks gestation); (ii) differences in proportions of the 2.5th percentiles of each of these measurements evaluated separately at 24-28 and 32-36 weeks gestation; (iii) Z-score trajectories of HC, AC, FL and EFW as a function of gestational age and intervention; and (iv) prevalence of small for gestational age (SGA) during the fetal period through birth as measured by WHO INTERGROWTH 21st standards.
Gestational age at birth | Up to 5 months (within 24 hours of birth, 3-5 months post randomization)
  In weeks, as continuous outcome, among all live births.
Preterm birth | Up to 5 months (within 24 hours of birth, 3-5 months post randomization)
  Preterm birth is defined as delivery of a living infant prior to 37 completed weeks of gestation.
WHO Non-severe Pneumonia | Up to 12 months after birth
  Cumulative incidence of WHO non-severe pneumonia (2014 definition and 2013 definition) during the first year of life. Cases of pneumonia are recorded whenever children present to HAPIN health facilities with respiratory symptoms.
WHO Severe Pneumonia | Up to 12 months after birth
  Cumulative incidence of WHO non-severe pneumonia (2014 definition and 2013 definition) during the first year of life. Cases of pneumonia are recorded whenever children present to HAPIN health facilities with respiratory symptoms.
Hospitalization for respiratory illness | Up to 12 months after birth
  Cumulative incidence of hospitalizations for a respiratory illness during the first year of life.
WHO Pocket Book Non-severe Pneumonia | Up to 12 months after birth
  Cumulative incidence of WHO non-severe pneumonia during the first year of life, as defined in the second edition of the "Pocket book of hospital care for children" (2013). Cases of pneumonia are recorded whenever children present to HAPIN health facilities with respiratory symptoms.
WHO Pocket Book Severe Pneumonia | Up to 12 months after birth
  Cumulative incidence of WHO severe pneumonia during the first year of life, as defined in the second edition of the "Pocket book of hospital care for children" (2013). Cases of pneumonia are recorded whenever children present to HAPIN health facilities with respiratory symptoms.
Hypoxemic Pneumonia | Up to 12 months after birth
  Cumulative incidence of hypoxemic pneumonia during the first year of life. Cases of pneumonia are recorded whenever children present to HAPIN health facilities with respiratory symptoms.
Ultrasound or Radiograph Pneumonia | Up to 12 months after birth
  Cumulative incidence of lung ultrasound or chest radiograph pneumonia during the first year of life. Cases of pneumonia are recorded whenever children present to HAPIN health facilities with respiratory symptoms.
Change in Brachial artery reactivity testing (BART) | Baseline, 18 months post-randomization
  Brachial artery reactivity testing (BART) measures endothelial function via flow-mediated dilatation to reactive hyperemia following the release of arm blood-flow occlusion. In this test, baseline artery diameter is measured, then a blood pressure cuff is inflated to induce distal arm ischemia for 5 minutes and after releasing the pressure, the post-occlusion brachial artery diameter is measured. The ratio of post- to pre-occlusion artery diameter represents endothelial function where lower values indicate worse endothelial function. (Peru only)
Change in Carotid intima-media thickness (CIMT) | Baseline, 18 months post-randomization, and when child is 24 months of age
  The carotid intima-media thickness test (CIMT) is used to determine the extent of carotid atherosclerotic vascular disease. The test measures the thickness of the inner two layers of the carotid artery and can detect plaque build up prior to physical symptoms being experienced. The carotid ultrasound will be performed with a portable ultrasound by trained sonographers.
Change in St. George Respiratory Questionnaire (SGRQ) Score | Baseline, 18 months post-randomization
  Adult respiratory health and well-being will be assessed with the St. George Respiratory Questionnaire (SGRQ). The SGRQ measures impaired health and perceived well-being among individuals with chronic airway disease. The SGRQ has sections assessing symptoms, activities that cause breathlessness or are limited because of breathlessness, and the impacts of respiratory problems on employment, sense of control of health, panic, stigmatization, medication use, side effects of therapies, expectations for health and disturbances of daily life. The questionnaire includes multiple choice, true/false and open-ended questions.
Change in Short Form 36 Survey (SF-36) Score | Baseline, 18 months post-randomization
  The Short Form 36 survey (SF-36) is a standardized, preference-based 36 item questionnaire evaluating quality of life. The survey has 8 sections (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health). Possible scores range from 0 (lowest quality of life) to 100 (highest quality of life).
Change in Weight | Baseline, 3, 6, 9, 12 and 18 months post-randomization, and at 24, 36, 48 and 60 months of age of the child
  Weight will be measured in the pregnant women/new mothers, the older adult women, and the children. Weight is measured in kilograms (kg). Weight in pregnant women will be measured at baseline, 24-28 weeks gestation, and 32-36 weeks gestation, and in new mothers when the child is 24- and 36-months old. In older adult women, it will be measured at baseline, 3, 6, 9, 12 and 18 months post-randomization, and when the child is 24-months old. Weight in children will be measured at birth, and at 3, 6, 9, 12, 24, 36, 48 and 60 months of age.
Change in Body Mass Index (BMI) | Baseline, 3, 6, 9, 12 and 18 months post-randomization, and at 24, 36, 48 and 60 months of age of the child
  BMI will be calculated for the pregnant women, the older adult women, and the children. BMI is calculated as weight in kilograms divided by height in meters (m) squared (kg/m²). BMI in pregnant women will be calculated at baseline, 24-28 weeks gestation, and 32-36 weeks gestation, and in new mothers when the child is 24- and 36-months old. In older adult women, it will be calculated at baseline, 3, 6, 9, 12 and 18 months post-randomization, and when the child is 24-months old. Weight in children will be calculated at birth, and at 3, 6, 9, 12, 24, 36, 48 and 60 months of age.
Change in Height | Baseline, 3, 6, 9, 12 and 18 months post-randomization, and at 24 months of age of the child
  Height in women will be measured in centimeters. Height in pregnant women will be measured at baseline, 24-28 weeks gestation, and 32-36 weeks gestation, and in new mothers when the child is 24- and 36-months old. In older adult women, it will be measured at baseline, 3, 6, 9, 12 and 18 months post-randomization, and when the child is 24-months old. This measurement will be used to compute the body mass index.
Change in Urinary Biomarkers | Baseline, 3, 6, 9, 12 and 18 months post-randomization, and 24 months of age of the child
  Multiple exposure biomarkers will be measured: 3-OH Cotinine, 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), levoglucosan, 8OH-deoxyguanosine (8OHdG), and Volatile Organic Chemicals (VOC) metabolites. Exposure biomarkers (especially for children whose urine may be limited) will be prioritized as follows: polycyclic aromatic hydrocarbon (PAH) biomarkers, levoglucosan, volatile organic chemicals (VOC) biomarkers, heavy metals, and tobacco-related biomarkers. Urinary biomarkers will be measured in pregnant women at baseline, 24-28 weeks gestation, and 32-36 weeks gestation, and in new mothers when the child is 24-months old. Biomarkers will be measured in older adult women at baseline, 3, 6, 9, 12 and 18 months post-randomization. Biomarkers will be measured in children at 3, 6, 12 and 24 months of age.
Change in Dried Blood Spot (DBS) Biomarkers | Baseline, 3, 6, 9, 12 and 18 months post-randomization, and at 24 months of age of the child
  The main biomarkers to be measured from the dried blood spots is: inflammation markers, endothelial markers of cardiovascular disease, oxidative stress markers, Hb, HbA1C, tumor-associated antigen antibodies, cytochrome P450, p53 tumor-associated antigen (TAA), lipids, metabolomics, MiRNA, heavy metals. DBS biomarkers will be measured in pregnant women at baseline, 24-28 weeks gestation, and 32-36 weeks gestation, and in new mothers when the child is 24-months old. DBS biomarkers will be measured in older adult women at baseline, 3, 6, 9, 12 and 18 months post-randomization. DBS biomarkers will be measured in children at 3, 6, 12 and 24 months of age.
Child Lung Function | 36, 48 and 60 months of age
  Lung function measurements will be made using the forced oscillation technique (FOT) with the Tremoflo C-100 device with disposable mouthpieces. FOT is a technique that can identify early changes in the airways. The FOT device measures the relationship between externally applied pressure waves and the resulting air flow to measure respiratory impedance. Values produced at high frequencies correspond to the proximal and large airways, and values produced at low frequencies correspond to distal and small airways. This measurement will be conducted in children in Guatemala.
Death | Up to Study Exit (up to 60 months of age of child)
  Death of all participants will be documented

OTHER OUTCOMES:
Change in fine particulate matter (PM2.5) exposure | Baseline, 3, 5, 9, 12 and 18 months post-randomization, and at 24, 36, 48, 60 months of age of the child
  Personal monitoring equipment will be used to assess exposure to fine particulate matter (PM2.5) over a 24-hour period in intervention and control participants (pregnant women, older adult women, and children). Exposure for pregnant women will be measured at baseline, 24-28 weeks gestation, 32-36 weeks gestation, and 24 months after delivery. Exposure in the child will be measured at 3, 6, 12, 24, 36, 48 and 60 months of age. Exposure in the older adult women will be measured at baseline, 3, 6, 12 and 18 months post-randomization, and at 24 months after delivery. Additionally, PM2.5 in the home will be measured 6 months, 12 months and 24 months after delivery of the child.
Change in Carbon monoxide (CO) exposure | Baseline, 3, 5, 9, 12 and 18 months post-randomization, and at 24, 36, 48, 60 months of age of the child
  Personal monitoring equipment will be used to assess exposure to carbon monoxide (CO) over a 24-hour period in intervention and control participants (pregnant women, older adult women, and children). Exposure for pregnant women will be measured at baseline, 24-28 weeks gestation, 32-36 weeks gestation, and 24 months after delivery. Children will be measured up to 12 months after delivery, and at 24, 36, 48 and 60 months of age. Older adult women will be measured up to 12 months after delivery, and at 24 months after delivery. Additionally, CO in the home will be measured 6 months, 12 months and 24 months after delivery of the child.
Change in Black carbon (BC) exposure | Baseline, 3, 5, 9, 12 and 18 months post-randomization, and at 24, 36, 48, 60 months of age of the child
  Personal monitoring equipment will be used to assess exposure to black carbon (BC) over a 24-hour period in intervention and control participants (pregnant women, older adult women, and children). Exposure for pregnant women will be measured at baseline, 24-28 weeks gestation, 32-36 weeks gestation, and 24 months after delivery. Children will be measured up to 12 months after delivery, and at 24, 36, 48 and 60 months of age. Older adult women will be measured up to 12 months after delivery, and at 24 months after delivery. Additionally, BC in the home will be measured 6 months, 12 months and 24 months after delivery of the child.
Maternal Perceived Stress Scale (PSS) | 9 to 18 months post-randomization (3 to 12 months of age of the child)
  The 10-item Cohen's Perceived Stress Scale (PPS) assesses the way an individual appraises their life events as stressful (e.g., "In the last month, how often have you felt difficulties were piling up so high that you could not overcome them?") (Cohen, 1983). Likert-level responses ranged from 0 (never) to 4 (very often), meaning a high PPS score would result in a high level of perceived stress. A Spanish language PPS created and tested and found to be valid and reliable (Vallijo et al., 2018).
Maternal death | Pregnancy through 42 days post-partum
  Death of a woman while pregnant or within 42 days of termination of pregnancy irrespective of the duration and site of the pregnancy.
Spontaneous abortion | Baseline through 20 weeks gestation
  Fetal death before 19 weeks 6 days.
Early preterm birth | Birth
  Births at less than 34 weeks completed gestation, among all live births.
Preterm delivery | Birth
  Including preterm birth and stillbirth.
Stillbirth | Up to birth
  Any fetal deaths occurring at or after 20 weeks' gestation OR indicated on Serious Adverse Event form OR on Pregnant Woman Medical History form OR on verbal autopsy form.
Neonatal death | Birth through 28 days
  Death between birth and 28 days.
Change in Child Blood Pressure | 48 and 60 months of age
  Blood pressure will be assessed in the children using automatic sphygmomanometers (OMRON HEM-907XL; Osaka, Japan). The study team will use the procedures adapted from previously validated methods and cardiovascular outcome studies, following recommendations for the American Heart Association and the European Society of Hypertension.
Change in Messenger Ribonucleic Acid (mRNA) Expression and microRNA in Older Adult Women | Baseline, 18 months post-randomization
  Two buccal cell scrapes will be collected by gently scraping the buccal mucosa on both sides of the mouth with a small plastic collection spoon. Nasal turbinate brush samples can be collected using a soft cytobrush on each turbinate. Collection is gentle and causes no discomfort to study participants. Both samples will be processed in the laboratory according to procedures detailed in the protocol. This will occur in the older adult women in an NCI substudy.
Change in Microbiome Operational Taxonomic Units (OTUs) in Older Adult Women | Baseline, 18 months post-randomization
  For the oral rinse, participants will vigorously rinse their mouth and the rinsates are collected in a centrifuge tube. The tube is centrifuged and the pellet and supernatant are removed to separate cryovials, labeled and frozen. This will occur in the older adult women in an NCI substudy.
Change in Epigenetics (DNA methylation) in Older Adult Women | Baseline, 18 months post-randomization
  Two buccal cell scrapes will be collected by gently scraping the buccal mucosa on both sides of the mouth with a small plastic collection spoon. A 5-mL venous blood sample will be collected in an ethylenediaminetetraacetic acid (EDTA) vacutainer tube by standard clinical venipuncture of a cubital vein. Both samples will be transported and processed in the laboratory according to procedures detailed in the protocol. This will occur in the older adult women in an NCI substudy.
Change in Metabolomics and MicroRNA in Older Adult Women | Baseline, 18 months post-randomization
  A 5-mL venous blood sample will be collected in an EDTA vacutainer tube by standard clinical venipuncture of a cubital vein. The sample will be transported and processed in the laboratory according to procedures detailed in the protocol. This will occur in the older adult women in an NCI substudy.
Household food insecurity | Baseline, 18 months post-randomization
  Household food insecurity will be measured using the Food Insecurity Experience Scale (FIES), developed and validated by the Food and Agriculture Organization (FAO). The FIES module includes eight questions, each with yes/no response options, on the household's access to adequate food, and is intended to measure three domains of food insecurity: uncertainty/anxiety, food quantity, and food quality. Each question takes values of 0/1, which are summed for a possible total score of 0-8.
Dietary diversity - women | Baseline to 18 months post-randomization
  Dietary diversity for women will be measured using the Minimum Dietary Diversity - Women (MDD-W) questionnaire from the FAO and FHI 360, which uses an open recall format to collect data on foods and beverages consumed by the respondent during the previous day and night. Responses will be categorized into ten food groups and women who report consuming five or more out of ten food groups will be categorized as achieving minimum dietary diversity.
Dietary diversity - infants | 9, 12, 15 and 18 months post-randomization (3, 6, 9, and 12 months of age), and 24, 36, 48 and 60 months of age
  Minimum dietary diversity for children will be measured using the World Health Organization (WHO) infant and young child feeding questionnaire. The questionnaire uses a combination of open and closed recall and asks caregivers to report on foods and beverages consumed by the infant or young child during the previous day and night. Responses will be categorized into eight food groups and infants who consumed five or more out of ten eight food groups will be categorized as achieving minimum dietary diversity.
Hemoglobin (Hb) concentration / anemia - women | Baseline, 3 and 5 months post-randomization
  Hb will be measured from a single drop of capillary blood obtained via finger prick, using the HemoCue® Hb 201system (HemoCue® AB) point-of-care device
Hemoglobin (Hb) concentration / anemia - infants | 12 and 18 months post-randomization (6 and 12 months of age)
  Hb will be measured from a single drop of capillary blood obtained via finger prick, using the HemoCue® Hb 201system (HemoCue® AB) point-of-care device

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clasen, PhD, Principal Investigator — Emory University; Jennifer Peel, PhD, Principal Investigator — Colorado State University; William Checkley, MD PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (4):
- Universidad del Valle de Guatemala, Guatemala City, Departamento de Guatemala, Guatemala
- Sri Ramachandra Institute of Higher Education and Research, Chennai, Tamil Nadu, India
- Puno Global Non-Communicable Disease Research Site, School of Medicine, Johns Hopkins University, Puno, Peru
- Rwanda Research Site, London School of Hygiene and Tropical Medicine, University of Liverpool, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearns KA, Naeher LP, McCracken JP, Boyd Barr D, Saikawa E, Hengstermann M, Mollinedo E, Panuwet P, Yakimavets V, Lee GE, Thompson LM. Estimating personal exposures to household air pollution and plastic garbage burning among adolescent girls in Jalapa, Guatemala. Chemosphere. 2024 Jan;348:140705. doi: 10.1016/j.chemosphere.2023.140705. Epub 2023 Nov 17. PMID 37981014
- [Background] Younger A, Ye W, Alkon A, Harknett K, Kirby MA, Elon L, Lovvorn AE, Wang J, Diaz-Artiga A, McCracken JP, Castanaza Gonzalez A, Alarcon LM, Mukeshimana A, Rosa G, Chiang M, Balakrishnan K, Garg SS, Pillarisetti A, Piedrahita R, Johnson MA, Craik R, Papageorghiou AT, Toenjes A, Williams KN, Underhill LJ, Hartinger SM, Nicolaou L, Chang HH, Naeher LP, Rosenthal J, Checkley W, Peel JL, Clasen TF, Thompson LM; Household Air Pollution Intervention Network (HAPIN) Investigators. Effects of a liquefied petroleum gas stove intervention on stillbirth, congenital anomalies and neonatal mortality: A multi-country household air pollution intervention network trial. Environ Pollut. 2024 Mar 15;345:123414. doi: 10.1016/j.envpol.2024.123414. Epub 2024 Jan 27. PMID 38286258
- [Background] Pillarisetti A, Ye W, Balakrishnan K, Rosa G, Diaz-Artiga A, Underhill LJ, Steenland K, Peel JL, Kirby MA, McCracken J, Waller L, Chang H, Wang J, Dusabimana E, Ndagijimana F, Sambandam S, Mukhopadhyay K, Kearns KA, Campbell D, Kremer J, Rosenthal J, Ghosh A, Clark M, Checkley W, Clasen T, Naeher L, Piedrahita R, Johnson M. Post-birth exposure contrasts for children during the Household Air Pollution Intervention Network randomized controlled trial. medRxiv [Preprint]. 2023 Jul 6:2023.07.04.23292226. doi: 10.1101/2023.07.04.23292226. PMID 37461598
- [Background] Simkovich SM, Hossen S, McCollum ED, Toenjes AK, McCracken JP, Thompson LM, Castanaza A, Diaz A, Rosa G, Kirby MA, Mukeshimana A, Myers R, Lenzen PM, Craik R, Jabbarzadeh S, Elon L, Garg SS, Balakrishnan K, Thangavel G, Peel JL, Clasen TF, Davila-Roman VG, Papageorghiou AT, de las Fuentes L, Checkley W; HAPIN Investigators. Lung Ultrasound Protocol and Quality Control of Image Interpretation Using an Adjudication Panel in the Household Air Pollution Intervention Network (HAPIN) Trial. Ultrasound Med Biol. 2023 May;49(5):1194-1201. doi: 10.1016/j.ultrasmedbio.2023.01.005. Epub 2023 Feb 19. PMID 36801180
- [Background] Williams KN, Quinn A, North H, Wang J, Pillarisetti A, Thompson LM, Diaz-Artiga A, Balakrishnan K, Thangavel G, Rosa G, Ndagijimana F, Underhill LJ, Kirby MA, Puzzolo E, Hossen S, Waller LA, Peel JL, Rosenthal JP, Clasen TF, Harvey SA, Checkley W; HAPIN Investigators. Fidelity and adherence to a liquefied petroleum gas stove and fuel intervention: The multi-country Household Air Pollution Intervention Network (HAPIN) trial. Environ Int. 2023 Sep;179:108160. doi: 10.1016/j.envint.2023.108160. Epub 2023 Aug 19. PMID 37660633
- [Background] Younger A, Alkon A, Harknett K, Kirby MA, Elon L, Lovvorn AE, Wang J, Ye W, Diaz-Artiga A, McCracken JP, Castanaza Gonzalez A, Monroy Alarcon L, Mukeshimana A, Rosa G, Chiang M, Balakrishnan K, Garg SS, Pillarisetti A, Piedrahita R, Johnson M, Craik R, Papageorghiou AT, Toenjes A, Quinn A, Williams KN, Underhill L, Chang HH, Naeher LP, Rosenthal J, Checkley W, Peel JL, Clasen TF, Thompson LM; HAPIN investigators. Effects of a LPG stove and fuel intervention on adverse maternal outcomes: A multi-country randomized controlled trial conducted by the Household Air Pollution Intervention Network (HAPIN). Environ Int. 2023 Aug;178:108059. doi: 10.1016/j.envint.2023.108059. Epub 2023 Jun 28. PMID 37413928
- [Background] Checkley W, Hossen S, Rosa G, Thompson LM, McCracken JP, Diaz-Artiga A, Balakrishnan K, Simkovich SM, Underhill LJ, Nicolaou L, Hartinger SM, Davila-Roman VG, Kirby MA, Clasen TF, Rosenthal J, Peel JL, On Behalf Of Household Air Pollution Intervention Network Hapin Investigators. Facing the Realities of Pragmatic Design Choices in Environmental Health Studies: Experiences from the Household Air Pollution Intervention Network Trial. Int J Environ Res Public Health. 2022 Mar 23;19(7):3790. doi: 10.3390/ijerph19073790. PMID 35409475
- [Background] Hennessee I, Kirby MA, Misago X, Mupfasoni J, Clasen T, Kitron U, Rosenthal JP, Hakizimana E. Assessing the Effects of Cooking Fuels on Anopheles Mosquito Behavior: An Experimental Study in Rural Rwanda. Am J Trop Med Hyg. 2022 Feb 21;106(4):1196-1208. doi: 10.4269/ajtmh.21-0997. Print 2022 Apr 6. PMID 35189594
- [Background] Johnson M, Pillarisetti A, Piedrahita R, Balakrishnan K, Peel JL, Steenland K, Underhill LJ, Rosa G, Kirby MA, Diaz-Artiga A, McCracken J, Clark ML, Waller L, Chang HH, Wang J, Dusabimana E, Ndagijimana F, Sambandam S, Mukhopadhyay K, Kearns KA, Campbell D, Kremer J, Rosenthal JP, Checkley W, Clasen T, Naeher L; the Household Air Pollution Intervention Network (HAPIN) Trial Investigators. Exposure Contrasts of Pregnant Women during the Household Air Pollution Intervention Network Randomized Controlled Trial. Environ Health Perspect. 2022 Sep;130(9):97005. doi: 10.1289/EHP10295. Epub 2022 Sep 16. PMID 36112539
- [Background] Kaufman JD. Invited Perspective: A Critical Part of a Real-World Environmental Health Trial Is to Demonstrate That the Intervention Reduced Exposure. Environ Health Perspect. 2022 Sep;130(9):91304. doi: 10.1289/EHP11697. Epub 2022 Sep 16. No abstract available. PMID 36112540
- [Background] Nicolaou L, Underhill L, Hossen S, Simkovich S, Thangavel G, Rosa G, McCracken JP, Davila-Roman V, de las Fuentes L, Quinn AK, Clark M, Diaz A, Pillarisetti A, Steenland K, Waller LA, Jabbarzadeh S, Peel JL, Checkley W; HAPIN Investigators. Cross-sectional analysis of the association between personal exposure to household air pollution and blood pressure in adult women: Evidence from the multi-country Household Air Pollution Intervention Network (HAPIN) trial. Environ Res. 2022 Nov;214(Pt 4):114121. doi: 10.1016/j.envres.2022.114121. Epub 2022 Aug 24. PMID 36029836
- [Background] Rajamani KD, Sambandam S, Mukhopadhyay K, Puttaswamy N, Thangavel G, Natesan D, Ramasamy R, Sendhil S, Natarajan A, Aravindalochan V, Pillarisetti A, Johnson M, Rosenthal J, Steenland K, Piedhrahita R, Peel J, Clark ML, Boyd Barr D, Rajkumar S, Young B, Jabbarzadeh S, Rosa G, Kirby M, Underhill LJ, Diaz-Artiga A, Lovvorn A, Checkley W, Clasen T, Balakrishnan K. Visualizing Field Data Collection Procedures of Exposure and Biomarker Assessments for the Household Air Pollution Intervention Network Trial in India. J Vis Exp. 2022 Dec 23;(190). doi: 10.3791/64144. PMID 36622010
- [Background] Ye W, Thangavel G, Pillarisetti A, Steenland K, Peel JL, Balakrishnan K, Jabbarzadeh S, Checkley W, Clasen T; HAPIN Investigators. Association between personal exposure to household air pollution and gestational blood pressure among women using solid cooking fuels in rural Tamil Nadu, India. Environ Res. 2022 May 15;208:112756. doi: 10.1016/j.envres.2022.112756. Epub 2022 Jan 20. PMID 35065931
- [Background] Ye W, Steenland K, Quinn A, Liao J, Balakrishnan K, Rosa G, Ndagijimana F, Ntivuguruzwa JD, Thompson LM, McCracken JP, Diaz-Artiga A, Rosenthal JP, Papageorghiou A, Davila-Roman VG, Pillarisetti A, Johnson M, Wang J, Nicolaou L, Checkley W, Peel JL, Clasen TF; Household Air Pollution Intervention Network (HAPIN) trial Investigators. Effects of a Liquefied Petroleum Gas Stove Intervention on Gestational Blood Pressure: Intention-to-Treat and Exposure-Response Findings From the HAPIN Trial. Hypertension. 2022 Aug;79(8):1887-1898. doi: 10.1161/HYPERTENSIONAHA.122.19362. Epub 2022 Jun 16. PMID 35708015
- [Background] Davila-Roman VG, Toenjes AK, Meyers RM, Lenzen PM, Simkovich SM, Herrera P, Fung E, Papageorghiou AT, Craik R, McCracken JP, Thompson LM, Balakrishnan K, Rosa G, Peel J, Clasen TF, Hossen S, Checkley W, de las Fuentes L; HAPIN Investigators. Ultrasound Core Laboratory for the Household Air Pollution Intervention Network Trial: Standardized Training and Image Management for Field Studies Using Portable Ultrasound in Fetal, Lung, and Vascular Evaluations. Ultrasound Med Biol. 2021 Jun;47(6):1506-1513. doi: 10.1016/j.ultrasmedbio.2021.02.015. Epub 2021 Apr 1. PMID 33812692
- [Background] Hengstermann M, Diaz-Artiga A, Otzoy-Sucuc R, Laura Maria Ruiz-Aguilar A, Thompson LM; HAPIN Investigators. Developing Visual Messages to Support Liquefied Petroleum Gas Use in Intervention Homes in the Household Air Pollution Intervention Network (HAPIN) Trial in Rural Guatemala. Health Educ Behav. 2021 Oct;48(5):651-669. doi: 10.1177/1090198121996280. Epub 2021 Mar 18. PMID 33733893
- [Background] Liao J, Kirby MA, Pillarisetti A, Piedrahita R, Balakrishnan K, Sambandam S, Mukhopadhyay K, Ye W, Rosa G, Majorin F, Dusabimana E, Ndagijimana F, McCracken JP, Mollinedo E, de Leon O, Diaz-Artiga A, Thompson LM, Kearns KA, Naeher L, Rosenthal J, Clark ML, Steenland K, Waller LA, Checkley W, Peel JL, Clasen T, Johnson M; HAPIN Investigators. LPG stove and fuel intervention among pregnant women reduce fine particle air pollution exposures in three countries: Pilot results from the HAPIN trial. Environ Pollut. 2021 Dec 15;291:118198. doi: 10.1016/j.envpol.2021.118198. Epub 2021 Sep 21. PMID 34740288
- [Background] Quinn AK, Williams KN, Thompson LM, Harvey SA, Piedrahita R, Wang J, Quinn C, Pillarisetti A, McCracken JP, Rosenthal JP, Kirby MA, Diaz Artiga A, Thangavel G, Rosa G, Miranda JJ, Checkley W, Peel JL, Clasen TF. Fidelity and Adherence to a Liquefied Petroleum Gas Stove and Fuel Intervention during Gestation: The Multi-Country Household Air Pollution Intervention Network (HAPIN) Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Nov 29;18(23):12592. doi: 10.3390/ijerph182312592. PMID 34886324
- [Background] Simkovich SM, Underhill LJ, Kirby MA, Crocker ME, Goodman D, McCracken JP, Thompson LM, Diaz-Artiga A, Castanaza-Gonzalez A, Garg SS, Balakrishnan K, Thangavel G, Rosa G, Peel JL, Clasen TF, McCollum ED, Checkley W; HAPIN Investigators. Resources and Geographic Access to Care for Severe Pediatric Pneumonia in Four Resource-limited Settings. Am J Respir Crit Care Med. 2022 Jan 15;205(2):183-197. doi: 10.1164/rccm.202104-1013OC. PMID 34662531
- [Background] Simkovich SM, Thompson LM, Clark ML, Balakrishnan K, Bussalleu A, Checkley W, Clasen T, Davila-Roman VG, Diaz-Artiga A, Dusabimana E, de las Fuentes L, Harvey S, Kirby MA, Lovvorn A, McCollum ED, Mollinedo EE, Peel JL, Quinn A, Rosa G, Underhill LJ, Williams KN, Young BN, Rosenthal J; HAPIN Investigators. A risk assessment tool for resumption of research activities during the COVID-19 pandemic for field trials in low resource settings. BMC Med Res Methodol. 2021 Apr 12;21(1):68. doi: 10.1186/s12874-021-01232-x. PMID 33845785
- [Background] Barr DB, Puttaswamy N, Jaacks LM, Steenland K, Rajkumar S, Gupton S, Ryan PB, Balakrishnan K, Peel JL, Checkley W, Clasen T, Clark ML; (HAPIN Investigative Team). Design and Rationale of the Biomarker Center of the Household Air Pollution Intervention Network (HAPIN) Trial. Environ Health Perspect. 2020 Apr;128(4):47010. doi: 10.1289/EHP5751. Epub 2020 Apr 29. PMID 32347765
- [Background] Burrowes VJ, Piedrahita R, Pillarisetti A, Underhill LJ, Fandino-Del-Rio M, Johnson M, Kephart JL, Hartinger SM, Steenland K, Naeher L, Kearns K, Peel JL, Clark ML, Checkley W; HAPIN Investigators. Comparison of next-generation portable pollution monitors to measure exposure to PM2.5 from household air pollution in Puno, Peru. Indoor Air. 2020 May;30(3):445-458. doi: 10.1111/ina.12638. Epub 2020 Jan 23. PMID 31885107
- [Background] Clasen T, Checkley W, Peel JL, Balakrishnan K, McCracken JP, Rosa G, Thompson LM, Barr DB, Clark ML, Johnson MA, Waller LA, Jaacks LM, Steenland K, Miranda JJ, Chang HH, Kim DY, McCollum ED, Davila-Roman VG, Papageorghiou A, Rosenthal JP; HAPIN Investigators. Design and Rationale of the HAPIN Study: A Multicountry Randomized Controlled Trial to Assess the Effect of Liquefied Petroleum Gas Stove and Continuous Fuel Distribution. Environ Health Perspect. 2020 Apr;128(4):47008. doi: 10.1289/EHP6407. Epub 2020 Apr 29. PMID 32347766
- [Background] Crocker ME, Hossen S, Goodman D, Simkovich SM, Kirby M, Thompson LM, Rosa G, Garg SS, Thangavel G, McCollum ED, Peel J, Clasen T, Checkley W; HAPIN Investigators. Effects of high altitude on respiratory rate and oxygen saturation reference values in healthy infants and children younger than 2 years in four countries: a cross-sectional study. Lancet Glob Health. 2020 Mar;8(3):e362-e373. doi: 10.1016/S2214-109X(19)30543-1. PMID 32087173
- [Background] Johnson MA, Steenland K, Piedrahita R, Clark ML, Pillarisetti A, Balakrishnan K, Peel JL, Naeher LP, Liao J, Wilson D, Sarnat J, Underhill LJ, Burrowes V, McCracken JP, Rosa G, Rosenthal J, Sambandam S, de Leon O, Kirby MA, Kearns K, Checkley W, Clasen T; HAPIN Investigators. Air Pollutant Exposure and Stove Use Assessment Methods for the Household Air Pollution Intervention Network (HAPIN) Trial. Environ Health Perspect. 2020 Apr;128(4):47009. doi: 10.1289/EHP6422. Epub 2020 Apr 29. PMID 32347764
- [Background] Puttaswamy N, Saidam S, Rajendran G, Arumugam K, Gupton S, Williams EW, Johnson CL, Panuwet P, Rajkumar S, Clark ML, Peel JL, Checkley W, Clasen T, Balakrishnan K, Barr DB. Cross-validation of biomonitoring methods for polycyclic aromatic hydrocarbon metabolites in human urine: Results from the formative phase of the Household Air Pollution Intervention Network (HAPIN) trial in India. J Chromatogr B Analyt Technol Biomed Life Sci. 2020 Oct 1;1154:122284. doi: 10.1016/j.jchromb.2020.122284. Epub 2020 Jul 29. PMID 32755815
- [Background] Sambandam S, Mukhopadhyay K, Sendhil S, Ye W, Pillarisetti A, Thangavel G, Natesan D, Ramasamy R, Natarajan A, Aravindalochanan V, Vinayagamoorthi A, Sivavadivel S, Uma Maheswari R, Balakrishnan L, Gayatri S, Nargunanathan S, Madhavan S, Puttaswamy N, Garg SS, Quinn A, Rosenthal J, Johnson M, Liao J, Steenland K, Piedhrahita R, Peel J, Checkley W, Clasen T, Balakrishnan K. Exposure contrasts associated with a liquefied petroleum gas (LPG) intervention at potential field sites for the multi-country household air pollution intervention network (HAPIN) trial in India: results from pilot phase activities in rural Tamil Nadu. BMC Public Health. 2020 Nov 26;20(1):1799. doi: 10.1186/s12889-020-09865-1. PMID 33243198
- [Background] Simkovich SM, Underhill LJ, Kirby MA, Goodman D, Crocker ME, Hossen S, McCracken JP, de Leon O, Thompson LM, Garg SS, Balakrishnan K, Thangavel G, Rosa G, Peel JL, Clasen TF, McCollum ED, Checkley W. Design and conduct of facility-based surveillance for severe childhood pneumonia in the Household Air Pollution Intervention Network (HAPIN) trial. ERJ Open Res. 2020 Mar 23;6(1):00308-2019. doi: 10.1183/23120541.00308-2019. eCollection 2020 Jan. PMID 32211438
- [Background] Williams KN, Thompson LM, Sakas Z, Hengstermann M, Quinn A, Diaz-Artiga A, Thangavel G, Puzzolo E, Rosa G, Balakrishnan K, Peel J, Checkley W, Clasen TF, Miranda JJ, Rosenthal JP, Harvey SA; Household Air Pollution Intervention Network (HAPIN) trial Investigators; HAPIN Investigators. Designing a comprehensive behaviour change intervention to promote and monitor exclusive use of liquefied petroleum gas stoves for the Household Air Pollution Intervention Network (HAPIN) trial. BMJ Open. 2020 Sep 29;10(9):e037761. doi: 10.1136/bmjopen-2020-037761. PMID 32994243
- [Background] Wilson DL, Williams KN, Pillarisetti A. 2020. An Integrated Sensor Data Logging, Survey, and Analytics Platform for Field Research and Its Application in HAPIN, a Multi-Center Household Energy Intervention Trial. Sustainability. 2020; 12 (5): 1805. doi:10.3390/su12051805.
- [Background] Goodman D, Crocker ME, Pervaiz F, McCollum ED, Steenland K, Simkovich SM, Miele CH, Hammitt LL, Herrera P, Zar HJ, Campbell H, Lanata CF, McCracken JP, Thompson LM, Rosa G, Kirby MA, Garg S, Thangavel G, Thanasekaraan V, Balakrishnan K, King C, Clasen T, Checkley W; HAPIN Investigators. Challenges in the diagnosis of paediatric pneumonia in intervention field trials: recommendations from a pneumonia field trial working group. Lancet Respir Med. 2019 Dec;7(12):1068-1083. doi: 10.1016/S2213-2600(19)30249-8. Epub 2019 Oct 4. PMID 31591066
- [Background] Liao J, McCracken JP, Piedrahita R, Thompson L, Mollinedo E, Canuz E, De Leon O, Diaz-Artiga A, Johnson M, Clark M, Pillarisetti A, Kearns K, Naeher L, Steenland K, Checkley W, Peel J, Clasen TF; HAPIN investigators. The use of bluetooth low energy Beacon systems to estimate indirect personal exposure to household air pollution. J Expo Sci Environ Epidemiol. 2020 Nov;30(6):990-1000. doi: 10.1038/s41370-019-0172-z. Epub 2019 Sep 26. PMID 31558836
- [Background] Quinn AK, Williams K, Thompson LM, Rosa G, Diaz-Artiga A, Thangavel G, Balakrishnan K, Miranda JJ, Rosenthal JP, Clasen TF, Harvey SA; HAPIN Investigators. Compensating control participants when the intervention is of significant value: experience in Guatemala, India, Peru and Rwanda. BMJ Glob Health. 2019 Aug 21;4(4):e001567. doi: 10.1136/bmjgh-2019-001567. eCollection 2019. PMID 31543990
- [Background] Steenland K, Pillarisetti A, Kirby M, Peel J, Clark M, Checkley W, Chang HH, Clasen T. Modeling the potential health benefits of lower household air pollution after a hypothetical liquified petroleum gas (LPG) cookstove intervention. Environ Int. 2018 Feb;111:71-79. doi: 10.1016/j.envint.2017.11.018. Epub 2017 Nov 26. PMID 29182949
- [Result] Checkley W, Thompson LM, Sinharoy SS, Hossen S, Moulton LH, Chang HH, Waller L, Steenland K, Rosa G, Mukeshimana A, Ndagijimana F, McCracken JP, Diaz-Artiga A, Balakrishnan K, Garg SS, Thangavel G, Aravindalochanan V, Hartinger SM, Chiang M, Kirby MA, Papageorghiou AT, Ramakrishnan U, Williams KN, Nicolaou L, Johnson M, Pillarisetti A, Rosenthal J, Underhill LJ, Wang J, Jabbarzadeh S, Chen Y, Davila-Roman VG, Naeher LP, McCollum ED, Peel JL, Clasen TF; HAPIN Investigators. Effects of Cooking with Liquefied Petroleum Gas or Biomass on Stunting in Infants. N Engl J Med. 2024 Jan 4;390(1):44-54. doi: 10.1056/NEJMoa2302687. PMID 38169489
- [Result] McCollum ED, McCracken JP, Kirby MA, Grajeda LM, Hossen S, Moulton LH, Simkovich SM, Goodman-Palmer D, Rosa G, Mukeshimana A, Balakrishnan K, Thangavel G, Garg SS, Castanaza A, Thompson LM, Diaz-Artiga A, Papageorghiou AT, Davila-Roman VG, Underhill LJ, Hartinger SM, Williams KN, Nicolaou L, Chang HH, Lovvorn AE, Rosenthal JP, Pillarisetti A, Ye W, Naeher LP, Johnson MA, Waller LA, Jabbarzadeh S, Wang J, Chen Y, Steenland K, Clasen TF, Peel JL, Checkley W; HAPIN Investigators. Liquefied Petroleum Gas or Biomass Cooking and Severe Infant Pneumonia. N Engl J Med. 2024 Jan 4;390(1):32-43. doi: 10.1056/NEJMoa2305681. PMID 38169488
- [Result] Balakrishnan K, Steenland K, Clasen T, Chang H, Johnson M, Pillarisetti A, Ye W, Naeher LP, Diaz-Artiga A, McCracken JP, Thompson LM, Rosa G, Kirby MA, Thangavel G, Sambandam S, Mukhopadhyay K, Puttaswamy N, Aravindalochanan V, Garg S, Ndagijimana F, Hartinger S, Underhill LJ, Kearns KA, Campbell D, Kremer J, Waller L, Jabbarzadeh S, Wang J, Chen Y, Rosenthal J, Quinn A, Papageorghiou AT, Ramakrishnan U, Howards PP, Checkley W, Peel JL; HAPIN Investigators. Exposure-response relationships for personal exposure to fine particulate matter (PM2.5), carbon monoxide, and black carbon and birthweight: an observational analysis of the multicountry Household Air Pollution Intervention Network (HAPIN) trial. Lancet Planet Health. 2023 May;7(5):e387-e396. doi: 10.1016/S2542-5196(23)00052-9. PMID 37164515
- [Result] Clasen TF, Chang HH, Thompson LM, Kirby MA, Balakrishnan K, Diaz-Artiga A, McCracken JP, Rosa G, Steenland K, Younger A, Aravindalochanan V, Barr DB, Castanaza A, Chen Y, Chiang M, Clark ML, Garg S, Hartinger S, Jabbarzadeh S, Johnson MA, Kim DY, Lovvorn AE, McCollum ED, Monroy L, Moulton LH, Mukeshimana A, Mukhopadhyay K, Naeher LP, Ndagijimana F, Papageorghiou A, Piedrahita R, Pillarisetti A, Puttaswamy N, Quinn A, Ramakrishnan U, Sambandam S, Sinharoy SS, Thangavel G, Underhill LJ, Waller LA, Wang J, Williams KN, Rosenthal JP, Checkley W, Peel JL; HAPIN Investigators. Liquefied Petroleum Gas or Biomass for Cooking and Effects on Birth Weight. N Engl J Med. 2022 Nov 10;387(19):1735-1746. doi: 10.1056/NEJMoa2206734. Epub 2022 Oct 10. PMID 36214599
- [Derived] Sivalogan K, Stein AD, Thompson LM, Wang J, Diaz-Artiga A, Aravindalochanan V, Jabbarzadeh S, Lovvorn AE, Ndagijimana F, Nicolaou L, Williams KN, Balakrishnan K, Peel JL, Checkley W, Clasen T, Sinharoy SS; HAPIN investigators paragraph sign. Provision of a liquefied petroleum gas cookstove and fuel during pregnancy and infancy and linear growth trajectories between birth and 12 months: Evidence from the multi-center Household Air Pollution Intervention Network (HAPIN) trial. PLOS Glob Public Health. 2025 Dec 31;5(12):e0004831. doi: 10.1371/journal.pgph.0004831. eCollection 2025. PMID 41474812
- [Derived] Pillarisetti A, Ye W, Peel JL, Chang H, Underhill LJ, Balakrishnan K, Diaz-Artiga A, McCracken JP, Rosa G, Thompson LM, Aravindalochanan V, Boyd Barr D, Chen Y, Chiang M, Clark ML, Davila-Roman V, Jabbarzadeh S, Johnson MA, Kirby MA, Lovvorn AE, Naeher LP, Ndagijimana F, Piedrahita R, Puttaswamy N, Waller LA, Wang J, Williams KN, Nicolaou L, Checkley W, Clasen TF, Rosenthal JP, Steenland K; HAPIN Investigators. Household air pollution and blood pressure among adult women participants of the Household Air Pollution Intervention Network Trial: An exposure-response analysis. Environ Res. 2025 Nov 15;285(Pt 5):122570. doi: 10.1016/j.envres.2025.122570. Epub 2025 Aug 12. PMID 40812702
- [Derived] Sivalogan K, Stein AD, Thompson LM, Wang J, Diaz-Artiga A, Aravindalochanan V, Jabbarzadeh S, Nicolaou L, Williams KN, Balakrishnan K, Peel JL, Checkley W, Clasen T, Sinharoy SS; HAPIN investigators. Provision of a liquefied petroleum gas cookstove and fuel during pregnancy and infancy and linear growth trajectories between birth and 12 months: evidence from the multi-center Household Air Pollution Intervention Network (HAPIN) trial. medRxiv [Preprint]. 2025 Jun 6:2025.06.05.25329099. doi: 10.1101/2025.06.05.25329099. PMID 40502604
- [Derived] Quinn A, Hengstermann M, Diaz-Artiga A, Pillarisetti A, Clark M, Ruiz-Aguilar L, Ndagijimana F, McCracken JP, Rosa G, Checkley W, Peel J, Clasen TF, Thompson L; HAPIN Investigators. Development of personal air pollution exposure report-back materials to Household Air Pollution Intervention Network (HAPIN) trial participants in Guatemala and Rwanda: a qualitative study. BMJ Glob Health. 2025 May 15;10(5):e017672. doi: 10.1136/bmjgh-2024-017672. PMID 40379277
- [Derived] Raheel H, Sinharoy S, Diaz-Artiga A, Garg SS, Pillarisetti A, Balakrishnan K, Chiang M, Lovvorn A, Kirby M, Ramakrishnan U, Jabbarzadeh S, Mukeshimana A, Johnson M, McCracken JP, Naeher LP, Rosa G, Wang J, Rosenthal J, Checkley W, Clasen TF, Peel JL, Thompson LM; Household Air Pollution Intervention Network (HAPIN) investigators. Effects of a liquefied petroleum gas stove and fuel intervention on head circumference and length at birth: A multi-country household air pollution intervention network (HAPIN) trial. Environ Int. 2025 Jan;195:109211. doi: 10.1016/j.envint.2024.109211. Epub 2024 Dec 24. PMID 39729872
- [Derived] Patil SS, Puttaswamy N, Cardenas A, Barr DB, Ghosh S, Balakrishnan K. Protocol for CARES-HAPIN: an ambidirectional cohort study on exposure to environmental tobacco smoke and risk of early childhood caries. BMJ Open. 2024 May 15;14(5):e083874. doi: 10.1136/bmjopen-2024-083874. PMID 38749682
- [Derived] Sivalogan K, Liang D, Accardi C, Diaz-Artiga A, Hu X, Mollinedo E, Ramakrishnan U, Teeny SN, Tran V, Clasen TF, Thompson LM, Sinharoy SS. Human Milk Composition Is Associated with Maternal Body Mass Index in a Cross-Sectional, Untargeted Metabolomics Analysis of Human Milk from Guatemalan Mothers. Curr Dev Nutr. 2024 Apr 10;8(5):102144. doi: 10.1016/j.cdnut.2024.102144. eCollection 2024 May. PMID 38726027
- [Derived] Checkley W, Thompson LM, Hossen S, Nicolaou L, Williams KN, Hartinger SM, Chiang M, Balakrishnan K, Garg SS, Thangavel G, Aravindalochanan V, Rosa G, Mukeshimana A, Ndagijimana F, McCracken JP, Diaz-Artiga A, Sinharoy SS, Waller L, Wang J, Jabbarzadeh S, Chen Y, Steenland K, Kirby MA, Ramakrishnan U, Johnson M, Pillarisetti A, McCollum ED, Craik R, Ohuma EO, Davila-Roman VG, de las Fuentes L, Simkovich SM, Peel JL, Clasen TF, Papageorghiou AT; Household Air Pollution Intervention Network (HAPIN) Investigators. Cooking with liquefied petroleum gas or biomass and fetal growth outcomes: a multi-country randomised controlled trial. Lancet Glob Health. 2024 May;12(5):e815-e825. doi: 10.1016/S2214-109X(24)00033-0. PMID 38614630
- [Derived] Simkovich SM, Thompson LM, Clark M, Balakrishnan K, Bussalleu A, Checkley W, Clasen T, Davila-Roman V, Diaz-Artiga A, de las Fuentes L, Harvey S, Kirby M, Lovvorn A, McCollum E, Peel J, Quinn A, Rosa G, Underhill L, Williams K, Young B, Rosenthal J. A Risk Assessment Tool for Resumption of Research Activities During the COVID-19 Pandemic. Res Sq [Preprint]. 2020 Nov 12:rs.3.rs-103997. doi: 10.21203/rs.3.rs-103997/v1. PMID 33200126

DOCUMENTS (8):
  • Statistical Analysis Plan: Stunting (Intention-to-treat) (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_006.pdf
  • Statistical Analysis Plan: Birthweight (Intention-to-treat and Exposure-Response) (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_000.pdf
  • Statistical Analysis Plan: Pneumonia (Intention-to-treat) (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_008.pdf
  • Statistical Analysis Plan: Anthropometry (Exposure-Response) (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_009.pdf
  • Statistical Analysis Plan: Blood Pressure in OAWs (Exposure-Response) (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_004.pdf
  • Statistical Analysis Plan: Blood Pressure in OAWs (Intention-to-treat) (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_005.pdf
  • Statistical Analysis Plan: Severe Pneumonia (Exposure-Response) (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/SAP_010.pdf
  • Informed Consent Form (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT02944682/ICF_001.pdf